CLINICAL TRIAL: NCT05212051
Title: A Randomized, Double-blind, Placebo-controlled, Phase II, Multicenter Study to Evaluate the Preliminary Efficacy, Safety, and Pharmacokinetics of Subcutaneous JS005 in Chinese Adult Patients With Active Ankylosing Spondylitis
Brief Title: Evaluate the Preliminary Efficacy, Safety, and PK of Subcutaneous JS005 in Chinese Adult Patients With Active AS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS005-003-II-AS
Record Dates: First submitted 2021-11-30; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Active Ankylosing Spondylitis

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator
Masking Description: Priticipant,Care provider and investigators are masked in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- JS005 150 mg (Experimental): 30 patients will be enrolled in this arm.
  Interventions: Biological: JS005
- Placebo 150 mg (Placebo Comparator): 10 patients will be enrolled in this arm.
  Interventions: Biological: Placebo
- JS005 300 mg (Experimental): 30 patients will be enrolled in this arm.
  Interventions: Biological: JS005
- Placebo 300 mg (Placebo Comparator): 10 patients will be enrolled in this arm.
  Interventions: Biological: Placebo
- JS005 450 mg (Experimental): 30 patients will be enrolled in this arm.
  Interventions: Biological: JS005
- Placebo 450 (Placebo Comparator): 10 patients will be enrolled in this arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: JS005 — 30 subjectes in JS005 150mg chort, JS005 300mg chort, and JS005 450mg chort receive JS005 150mg, JS005 300mg and JS005 450mg subcutaneous injection seperately at Week 0, 1, 2, and 3, and monthly dose starting at Week 4 (dosing in Week 4, 8, and 12).
  Other Names: Recombinant humanized anti-IL-17A monoclonal antibody injection
  Arms: JS005 150 mg; JS005 300 mg; JS005 450 mg
Biological: Placebo — 10 subjects in JS005 150mg chort, JS005 300mg chort, and JS005 450mgchort receive the placebo subcutaneous injection seperately at Week 0, 1, 2, and 3, and monthly dose starting at Week 4 (dosing in Week 4, 8, and 12).
  Arms: Placebo 150 mg; Placebo 300 mg; Placebo 450

SUMMARY:
The purpose of this study is to evaluate preliminary efficacy, safety pharmacokinetic (PK) characteristics, pharmacodynamics (PD) haracteristics and immunogenicity of JS005 at different doses in Chinese patients with active Ankylosing Spondylitis. Treatment difference of JS005 150mg,300mg,450mg vs. placebo in Chinese AS patients in terms of ASAS 20 response rate at Week 16 as well as safety profile will be provided by the study .

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. Approximately 120 patients who meet the eligibility criteria will be randomized to one of three treatment cohorts (JS005 150 mg, 300 mg, 450mg in a ratio of 1:1:1),then using secondary randomization method, 40 patients in each group will be randomized in a 3: 1 ratio to receive investigational product or placebo.

1. JS005 150mg Cohort: JS005 150 mg or placebo treatment(JS005:Placrbo=3:1) s.c. prefilled syringe (PFS) on Week 0, 1, 2, 3, 4,8 and 12
2. JS005 300mg Cohort: JS005 300 mg or placebo treatment(JS005:Placrbo=3:1) s.c. PFS on Week0, 1, 2 ,3, 4,8,and 12 3 .JS005 450mg Cohort: JS005 450 mg or placebo treatment(JS005:Placrbo=3:1) s.c. PFS on Week0, 1, 2 ,3, 4,8,and 12 Based on the clinical judgment of disease activity by the investigator and the patient, background medications, such as NSAIDs and DMARDs, may have been modified or added to treat signs and symptoms of AS from Week 16 on.

ELIGIBILITY:
Inclusion Criteria:

1. Have an established diagnosis of AS according to Modified New York criteria for AS in 1984, and active AS assessed by total BASDAI ≥ 4 (0-10 point scale) and spinal pain ≥ 4 （according to the 0-10 NRS scale ( BASDAI question #2) at baseline.
2. Voluntarily participate in this clinical trial and sign the informed consent form.
3. Male or female aged between 18 and 65 years (both inclusive) at the time of signing informed consent. Female subjects of childbearing age are required to have a confirmed negative result of urine and/or serum pregnancy test performed within 3 days before randomization and agree to use reliable contraceptive measures during the study; Male patients and their female partners of childbearing age must agree to use reliable contraception during the study.
4. Patients meet at least one of the following: 1) have an inadequate or ineffective response to NSAIDs, 2) have been intolerant to at least one dose of NSAIDs, 3) have contraindications to NSAIDs therapy. Inadequate or ineffective response to NSAIDs is defined as no remission after continuous treatment with standard doses of at least 2 NSAIDs for a total of no less than 4 weeks and no less than 2 weeks for each NSAID.
5. Patients regularly taking NSAIDs as part of their AS therapy are required to maintain a stable dose for at least 2 weeks prior to randomization.
6. Patients using tumor necrosis factor α (TNFα) inhibitors must have experienced an inadequate response to the standard treatment doses for at least 3 months, or have been intolerant to anti-TNFα agents.
7. Patients who have previously been on a TNFα inhibitor will be allowed entry into study after an appropriate wash-out period prior to randomization (e.g., washout periods of 4 weeks for etanercept, 8 weeks for infliximab, and 10 weeks for adalimumab, golimumab, and certolizumab, respectively).
8. Patients taking Methotrexate (MTX) (≤ 25 mg/week) or sulfasalazine (SSZ) ( ≤ 3 g/day) are allowed to continue their medication and must have taken it for at least 3 months and be on a stable dose for at least 4 weeks prior to randomization. Patients taking MTX need to take folic acid supplements.
9. Patients who are on conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs) other than MTX and sulfasalazine must discontinue the csDMARDs 4 weeks prior to randomization, except for leflunomide (LEF), which has to be discontinued for 8 weeks prior to randomization unless a cholestyramine washout has been performed.
10. Patients taking systemic corticosteroids have to be on a stable dose of ≤ 10 mg/day prednisone or equivalent for at least 2 weeks prior to randomization

Exclusion Criteria:

1. Patients with total ankylosis of the spine or imaging (X-ray) with the evidence of sacroiliitis with complete fusion of sacroiliac joints.
2. Previous exposure to JS005 or any other biologic drug directly targeting IL-17 or IL-17 receptors.
3. Have taken high potency analgesics (e.g., opiates of methadone, hydromorphone, morphine) within 2 weeks prior to randomization.
4. Previous treatment with any intra-articular injection (e.g., glucocorticoids) within 4 weeks prior to randomization.
5. Previous treatment with any biological immunomodulating agents other than the TNFα inhibitors.
6. Treatment with JAK inhibitor agents within 8 weeks prior to randomization and unwilling to discontinue during the study.
7. Patient unwilling to take folic acid/leucovorin to reduce MTX toxicity.
8. Has received any cell-depletion therapies including but not limited to anti-CD20 antibodies, or investigational agents (e.g., Campath, anti-CD4 , anti-CD5, anti-CD3, anti-CD19).
9. Previous treatment with traditional Chinese medicine or animal and plant extracts for AS within 4 weeks prior to randomization.
10. Use of any investigational agents and/or devices within 4 weeks prior to randomization or within 5 half-lives of the investigational drug, whichever is longer.
11. Females who are pregnant or lactating.
12. Chest imaging (e.g., x-ray or CT) with evidence of ongoing infectious or malignancy, obtained within 3 months prior to screening and evaluated by a qualified physician
13. Active systemic infections (other than the common cold) within 2 weeks prior to randomization.
14. Patients with other diseases other than ankylosing spondylitis that might confound the evaluation of the efficacy of JS005 therapy: such as chronic pain other than ankylosing spondylitis (such as fibromyalgia), inflammatory bowel disease, acute anterior uveitis, etc., within 6 weeks prior to randomization. However, patients with non-acute iritis and psoriasis that have been stable for 6 months or more can be included in this study.
15. Underlying metabolic, hematologic, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, or gastrointestinal conditions which in the opinion of the investigator immunocompromises the patient and/or places the patient at unacceptable risk in case of using immunomodulatory therapy.
16. Myocardial infarction, apoplexy, congestive heart failure (New York Heart Association status of class III or IV) within 6 months prior to screening; uncontrolled hypertension (≥ 160/95 mmHg) prior to randomization.
17. Patients with type 1 diabetes mellitus, or newly diagnosed or uncontrolled type 2 diabetes mellitus (e.g., HbA1C > 9.0%) within 6 months prior to screening.
18. Patients with active liver disease or hepatic insufficiency, with any of the following abnormalities in liver function tests at screening: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin > 1.5 × upper limit of normal.
19. History of renal injury, glomerulonephritis, or patient with only one kidney or glomerular filtration rate < 60 mL/(min · 1.73 m2 ) at screening.
20. Total white blood cell count < 3 × 109/L, or neutrophils < 1.5 × 109/L or absolute lymphocyte count < 0.5 × 109/L or hemoglobin < 8.5 g/dL or platelets < 100 × 109/L at screening.
21. History of ongoing chronic or recurrent infectious disease, or evidence of tuberculosis infection on tuberculosis screening (X. DOT-TB, QuantiFERON TB-Gold, T-SPOT) (see Section 8.3.4 for details).
22. Positive for human immunodeficiency virus antibody (Anti-HIV) at screening.
23. Positive for hepatitis C virus antibody (Anti-HCV) at screening.
24. HBV DNA is detected in patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at screening (the lower limit of quantitative detection refers to the reference value of each hospital.).
25. History of lymphoproliferative disease or malignancy within the past 5 years (except for basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 3 months, and carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been surgically removed ).
26. Previous or medical history of other significant concomitant diseases that, in the judgment of the investigator, participation would not be in the best interest of the patient. These include, but are not limited to, cardiovascular disorder, nephropathy, neurological disease (including demyelinating disease), active infectious disease, endocrine disease, gastrointestinal disease, hepatobiliary disease, metabolic disease, pulmonary disease, non-malignant lymphoproliferative disease, or other lymphatic diseases.
27. Surgery of the spine or joint or other major surgery (e.g., aneurysmectomy, gastric ligation) within 3 months prior to randomization or planned during the study.
28. History or evidence of ongoing alcohol or drug abuse within 6 months prior to randomization.
29. The patient has a history of systemic hypersensitivity to any biological agent, excluding injection site reactions.
30. Vaccination with a live vaccine (live attenuated vaccine*) and BCG vaccine within 12 weeks prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-11-02 (Estimated); Study Completion 2023-01-11 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | From week 0 to week 16
  The proportion of AS patients meeting the Assessment of Spondylo Arthritis international Society 20 (ASAS20) response criteria at the end of treatment Week 16.

SECONDARY OUTCOMES:
ASAS40 response criteria | From week 0 to week 16
  The proportion of patients meeting the ASAS40 response criteria at the end of treatment Week 16;
ASAS 5/6 response criteria | From week 0 to week 16
  The proportion of patients meeting the ASAS 5/6 response criteria at the end of treatment Week 16;
High-sensitivity C-reactive protein (hsCRP) | From week 0 to week 16
  The change from baseline in high-sensitivity C-reactive protein (hsCRP) at the end of treatment Week 16
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | From week 0 to week 16
  The change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at the end of treatment Week 16;
Bath Ankylosing Spondylitis Functional Index (BASFI) | From week 0 to week 16
  The change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at the end of treatment Week 16
Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) | From week 0 to week 16
  The change from baseline in Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) at the end of treatment Week 16
Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) | From week 0 to week 16
  The change from baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at the end of treatment Week 16
The proportion of patients meeting the ASAS partial remission criteria | From week 0 to week 16
  The proportion of patients meeting the ASAS partial remission criteria at the end of treatment Week 16
nkylosing Spondylitis Disease Activity Score (ASDAS-CRP) | From week 0 to week 16
  The change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) at the end of treatment Week 16;
The patient's global assessment of disease activity | From week 0 to week 16
  The change from baseline in the patient's global assessment of disease activity at the end of treatment Week 16
The patient's assessment of inflammatory back pain intensity | From week 0 to week 16
  The change from baseline in the patient's assessment of inflammatory back pain intensity at the end of treatment Week 16

OTHER OUTCOMES:
Pharmacokinetic endpoint | From baseline to week 24, Total 24 weeks
  Population pharmacokinetic analysis of plasma concentrations will be performed to explore the exposure of JS005 in patients and the influencing factors of exposure
Pharmacodynamic endpoint | From baseline to week 24, Total 24 weeks
  Concentrations and the changes of free and/or total IL-17 in serum before and after administration.
Immunogenicity endpoint | From baseline to week 24, Total 24 weeks
  Anti-drug antibody (ADA), for the ADA positive samples, it is necessary to test the titer and determine whether it is a neutralizing antibody (Nab).
Safety evaluation | From V1 to V12, Total 36 Weeks
  Safety evaluation includes AE monitoring, physical examination, vital signs, electrocardiograph (ECG), clinical laboratory tests (hematology, serum chemistry and urinalysis) throughout the study, recording the clinical manifestations, severity, occurrence time, end time, treatment measures and outcomes, and determining the correlation between AE and the investigational product.

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Shamen, Fujian
  - Sun Yat-sen Memorial Sun Yat-sen University City: Guangzhou, Guangzhou, Guangdong
  - Nanfang Hospital of Nandang Medical University, Guangzhou, Guangdong
  - Shantou University Medical Collge No.1 Affiliated Hospital, Shantou, Guangdong
  - Pking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Gudong
  - Tianjin Medical University General Hospital, Tianjin, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical college of HUST, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affilated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China medical University, Shengyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Chuanbei Meidical College Affiliated Hospital, Nanchong, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang